CLINICAL TRIAL: NCT03620071
Title: Intelligent Information Sharing: Advancing Teamwork in Complex Care
Brief Title: GoalKeeper: Intelligent Information Sharing for Children With Medical Complexity
Acronym: GoalKeeper
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Harvard University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R01CA204585-01 (NIH); 1R01CA204585-01 (NIH)
Record Dates: First submitted 2018-07-19; First posted 2018-08-08 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Childhood Cancer; Cerebral Palsy; Chronic Lung Disease; Congenital Heart Disease; Congenital Metabolic Disorder; Gastrostomy
Keywords: complex chronic condition; care coordination; shared decision making; health literacy
MeSH Terms: conditions — Neoplasms; Cerebral Palsy; Heart Defects, Congenital; Metabolism, Inborn Errors | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Receipt of a novel mobile-health tool, GoalKeeper Plus Standard Care
  Interventions: Other: GoalKeeper; Other: Standard Care
- Control (Experimental): Standard Care
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: GoalKeeper — Mobile-health communication tool for parents of children with medical complexity
  Arms: Intervention
Other: Standard Care — Standard Clinical Care

SUMMARY:
This proposal addresses the major challenge of improving health outcomes for children with cancer and other complex conditions, for whom the effectiveness of outpatient care depends on care coordination across a diverse group of caregivers that includes parents, community support organizations and pediatric care providers. The investigators have developed GoalKeeper, a prototype system for supporting care coordination across multiple care providers. The primary aim of the clinical trial is to assess the potential for this new system, GoalKeeper, to improve meaningful use of goal-centered care plans in the care of children with cancer and other complex chronic conditions.

DETAILED DESCRIPTION:
The overarching aim of the research is to improve care coordination and goal setting for children with medical complexity (CMC). Specific aims of the pilot clinical trail are as follows: (1) To assess the efficacy of GoalKeeper on goal-setting in the health care encounter. (2) To examine the roles of parent health literacy and parent activation in moderating the effect of the intervention.

Study Population: Stanford's Primary and Subspecialty Care Clinics at Stanford Children's Health will serve as the setting for study recruitment.

The pilot randomized controlled trial will enroll 60 parents of children with medical complexity and their health-care providers. Eligibility criteria for participants will be age 18 years or older, English-speaking, and (for parents) child<12 years old. Exclusion criteria are parent with known mental illness or neurocognitive impairment. A stepped wedge approach by provider will introduce families to GoalKeeper at different time points in the study. A pre-intervention period will occur at least 1 month before the trial start where clinical observations and baseline survey information will be obtained of each providers' practice.

Each family will be given training and 4-month access to the GoalKeeper application and participate in an exit interview at the end of study.

ELIGIBILITY:
Inclusion Criteria:

* Parent-child dyads and their medical provider
* Parent and provider age 18 years or older
* Parent English- or Spanish-speaking
* Child > age 12 months and <12 years old

Exclusion Criteria:

* Parent with known mental illness or neurocognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-03-17 (Actual)

PRIMARY OUTCOMES:
Change in Parent Perception of Goal-Centered Care questionnaire from Baseline to 1-Month Follow-up | Baseline and 1-Month Follow-up
  Parent perception of goal-centered care will be measured using a modified version of the "Patient Assessment of Chronic Illness Care, Goal-Setting Domain" questionnaire, using a scale of 1(Almost Never) to 5 (Almost Always) with higher values representing better goal-centered care.

SECONDARY OUTCOMES:
Count of parent participants with change in perception of goal-centered care from baseline to 3-Month Follow-up based on Investigator assessment. | Baseline and 3 month follow-up
  Change in perception in quality of goal-centered care will be assessed by Investigators based on parent baseline interviews and parent exit interviews.

OTHER OUTCOMES:
Change in parent perception of quality of shared decision making from baseline to 1 month | Baseline and 1-Month Follow-up
  Parent perception will be measured using the "National Survey of Children with Special Health Care Needs Shared Decision Making Domain," which includes 4 domain items each with a scale of 1 (never), 2 (sometimes), 3 (usually) or 4 (always). Positive SDM is defined as parent report of "usually" or "always" on all 4 items. Shared decision making refers to a communication process where parents and providers participate in decision making to reach treatment plan agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Lee M Sanders, MD, MPH, Principal Investigator — Associate Professor, Pediatrics
Locations (1):
- Stanford Children's Health, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lin JL, Clark CL, Halpern-Felsher B, Bennett PN, Assis-Hassid S, Amir O, Nunez YC, Cleary NM, Gehrmann S, Grosz BJ, Sanders LM. Parent Perspectives in Shared Decision-Making for Children With Medical Complexity. Acad Pediatr. 2020 Nov-Dec;20(8):1101-1108. doi: 10.1016/j.acap.2020.06.008. Epub 2020 Jun 12. PMID 32540424
- [Derived] Lin JL, Huber B, Amir O, Gehrmann S, Ramirez KS, Ochoa KM, Asch SM, Gajos KZ, Grosz BJ, Sanders LM. Barriers and Facilitators to the Implementation of Family-Centered Technology in Complex Care: Feasibility Study. J Med Internet Res. 2022 Aug 23;24(8):e30902. doi: 10.2196/30902. PMID 35998021